CLINICAL TRIAL: NCT02707198
Title: Prevention of Clostridium Difficile-associated Diarrhea by Daily Intake of Kefir
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study was not feasible to complete at study site
Sponsor: St. Luke's Hospital of Duluth (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: C. diff
Record Dates: First submitted 2015-12-30; First posted 2016-03-14 (Estimated); Results first posted 2022-05-19 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Clostridium Difficile Infection; Diarrhea
MeSH Terms: conditions — Clostridium Infections; Diarrhea | interventions — Kefir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A (No Intervention): Will receive prescribed antibiotics and will not receive kefir. Patients in this arm will be asked to record daily symptoms of diarrhea for up to 30 days post-discharge.
- Group B (Active Comparator): Will receive prescribed antibiotics and will receive kefir only during hospital stay. Patients in this arm will be asked to record daily symptoms of diarrhea for up to 30 days post-discharge.
  Interventions: Drug: kefir
- Group C (Active Comparator): Will receive prescribed antibiotics and will receive kefir during hospital stay and for the duration of the prescribed antibiotic regimen for up to a total of 30 days . Patients in this arm will be asked to record daily symptoms of diarrhea for up to 30 days post-discharge.
  Interventions: Drug: kefir

INTERVENTIONS:
Drug: kefir — 4 ounces of kefir 3 times a day, with or without food.
  Arms: Group B; Group C

SUMMARY:
This study is being conducted to investigate the potential benefits of probiotic intake for preventing antibiotic associated diarrhea and Clostridium difficile infection in patients undergoing a systemic antibiotic treatment. The primary research question is: can daily intake of kefir, a yogurt-like food containing probiotics, reduce the incidence of diarrhea and Clostridium difficile infection in patients during antibiotic treatment?

DETAILED DESCRIPTION:
Background and Significance

Clostridium difficile infections are of great concern for hospitals nationwide and C. difficile remains the most common nosocomial infection in North America. The majority of patients with C. difficile infection respond to orally administered metronidazole or vancomycin, but 5-30% of patients go on to develop recurrent infection and diarrhea, despite antibiotic treatments. The idea that gut microbiota influence susceptibility and recovery from disease is becoming more widely reported. Disruption of normal bacterial flora in the gut during systemic antibiotic use has been attributed to the uncontrolled growth of bacteria that are otherwise suppressed such as C. difficile. Even after an antibiotic regimen has concluded, restoration of the normal gut microbiota is thought to be paramount to interrupting the cycle of C. difficile infection. The idea of reintroducing normal microbial flora to patients with recurrent C. difficile infections has been the foundation upon which the use of probiotic agents, including fecal transplants, has been introduced. The use of probiotics to treat antibiotic-associated diarrhea, and specifically C. difficile infections, has been studied and successes have been reported, and in particular by our group. The emerging idea, however, is that probiotic consumption can be used to prevent the onset of a C. difficile infection, which requires further study. Meta-analyses have been conducted on previously reported data and ultimately conclude that the use of probiotics is safe and effective. However, there remains a need for a focused and controlled study assessing the efficacy of kefir consumption on the incidence of C. difficile infections at St. Luke's Hospital in Duluth, MN, and CHI Creighton University Medical Center in Omaha, NE. The data collected from this study have the potential to change clinical practice at not only our institutions, but at any hospital or institution that has a population of patients undergoing systemic antibiotic treatment.

Risk factors for persistent C. difficile infection include age greater than 65 years, poor nutritional status, recent abdominal surgery, prolonged hospitalization and recent stay in the ICU. The purpose of this study is to determine if administering a daily regimen of kefir to at-risk patients can reduce the incidence of C. difficile infections. Because treatment for C. difficile infections is difficult and expensive, and recurrent infections are common, a way to prevent these infections is of great interest. A preventive measure that reduces the incidence of diarrhea and C. difficile infections will clearly improve patient health, and will have a multi-fold impact on how patients are cared for while in the hospital as well as post-discharge. There is potential for cost-saving, as well, in the form of the direct cost of antibiotic treatments and prolonged hospital stays. Additionally, the cost in time and effort to prevent the spread of these infections will be reduced, as well, all of which ultimately improve patient care.

Preliminary Studies

Many studies have been published indicating a potential for probiotics as a prophylaxis against diarrhea associated with antibiotic use in humans. Additionally, a recent report in a rodent model suggests that kefir consumption concomitantly with antibiotic treatment may prevent the development of C. difficile-associated diarrhea. However, to our knowledge there have not been any studies published that have investigated the preventive effects of kefir consumption specifically related C. difficile infection in human patients. This protocol will serve as an initial study for a subset of at-risk patients and the data collected will provide guidance for future studies to include a more broad range of at-risk patients.

Research Design and Methods

Subjects

The study will include patients who have been prescribed a systemic antibiotic of any kind (administered by oral or parenteral route), but have not yet begun the treatment regimen. There will be three study groups:

* Group A: Patients receive antibiotics and receive no kefir
* Group B: Patients receive antibiotics and receive kefir during their hospital stay only
* Group C: Patients receive antibiotics and receive kefir following discharge for the duration of their antibiotic regimen, for a maximum of 30 days

All patients will receive a journal to track their kefir intake (if in Group C) and any loose stools or diarrhea for 30 days after their hospital stay. Additionally, all patients will receive a follow-up phone call 3-5 days after discharge from the hospital, and weekly thereafter for 30 days, to determine if diarrhea has occurred. All patients will be instructed to call their physician if symptoms of diarrhea occur. The aims of this study are to determine the incidence of antibiotic-associated diarrhea in each of the study groups as well as the presence of C. difficile in the stool of those patients that report having diarrhea.

Data Collection and Accrual Methods

Patients who meet inclusion criteria and consent to be part of the study will be assigned to one of the three study groups at random.

During the standard admissions interview, patients are asked about any allergies, including milk protein allergy. This type of allergy will exclude patients from participating in the study. Because kefir is 99% lactose free, lactose intolerance will not exclude individuals from participating. Per standard of care, a physical exam will be performed and a symptom-directed exam will be performed at any follow-up appointments, typically one month after discharge from the hospital.

Patients in study groups consuming kefir will receive an information card that includes the nutrition facts for a 4-ounce serving of kefir. Lifeway brand Kefir® will be used as it is widely available and comes in several palatable flavors. The probiotic content of Lifeway Kefir remains constant, regardless of flavor.

Patients in Group A will receive their prescribed antibiotics during their hospital stay and will not receive kefir. These patients will be instructed to not consume any yogurt, kefir, or other probiotic products during their hospital stay and for 30 days post-discharge.

Patients in Groups B and C will begin receiving kefir on the same day that their prescribed antibiotic regimen begins. Four ounces of kefir will be administered 3 times a day to patients enrolled on this study. A 4 oz. glass of kefir will be provided with every mealtray, and nursing staff at each of the participating institutions will administer the kefir to the patients. The amount of kefir consumed by the patient will be recorded by the nursing staff and entered in the electronic medical record. Four ounces is a standard serving of yogurt and is well-tolerated by patients. This serving size will help maintain ongoing live probiotic cultures in the individuals receiving kefir.

For patients in Group B, administration of kefir by the nursing staff will continue for the duration of the patients' hospital stay only. For patients in Group C, kefir will be prescribed at the same dose as given during their hospital stay (at least 4 ounces of kefir 3 times each day, not to exceed 12 ounces per day).

All patients will be given a journal in which they can record any symptoms of a C. difficile infection (i.e., diarrhea). Additionally, patients in Group C will record their kefir consumption on a daily basis. All patients will receive a follow-up phone call 3 days after their hospital discharge and weekly thereafter for 30 days (a total of 4 phone calls). Patients will be asked if they have had any incidence of diarrhea in order for nursing staff and physicians to assess if C. difficile infection has occurred.

All patients will be asked to contact their physician if they experience diarrhea after their hospital stay. These patients will be offered a fecal C. difficile test, as per standard of care. Any patient that has 3 or more watery stools in a 24 hour period and a positive C. difficile stool test will be considered as having a C. difficile infection. Stool collection and testing will be carried out per treatment guidelines. No further typing of C. difficile isolates will be performed on samples obtained as it is beyond the scope of this study.

Patients who develop a C. difficile infection during the study will be immediately treated per standard of care and will be considered treatment failures. However, these patients will be contacted for follow-up information pertinent to the study (i.e., duration of symptoms, and efficacy of standard treatment). Follow up contacts will be made via telephone; an initial call will be made 3 days post discharge from the hospital and patients will be contacted weekly thereafter for 30 days. During these phone calls, patients will be asked if they have any concerns or symptoms, specifically related to diarrhea.

If at any point during the hospitalization or during the follow-up timeframe a patient receiving kefir displays signs or symptoms of an invasive bacterial, yeast, or fungal infection, blood cultures and other cultures as deemed clinically appropriate (urine culture, sputum culture, wound culture, etc.) will be obtained. Signs and symptoms of an invasive infection include, but are not limited to, the following: fever, chills, elevated WBC concentration, elevated serum C-reactive protein (CRP) and/or procalcitonin levels, and hypotension.

If a suspected invasive infection occurs during the course of kefir administration, the following empiric treatment regimen will be considered:

• Intravenous administration of vancomycin plus piperacillin/tazobactam plus fluconazole

* Intravenous daptomycin will be used for patients with a previously documented vancomycin allergy
* An intravenous fluoroquinolone (ciprofloxacin or moxifloxacin) will be used for patients with a documented penicillin allergy
* Intravenous micafungin will be used for patients with a documented fluconazole allergy

Initial intake screening for inclusion in the kefir research study will include an evaluation of known allergies. Antibiotic therapy will be adjusted in accordance with identification of the causative organism(s) and corresponding antibiotic susceptibilities. Treatment duration will be determined based on standards of care for the clinical situation and the causative organism.

Data Analysis

The three treatment groups will be compared using logistic regression with covariates of study location, age, gender, antibiotic type and doses, hypoalbuminemia, and compromised immune system. Model selection based on the Akaike Information Criterion will be used to select covariates in final models. The treatment groups will also be compared without covariate adjustment. As needed, missing data will be handled using multiple imputation after assessment of missing at random considerations. Dependent and independent variables in planned analyses will be included in imputations along with any auxiliary variables thought to be potentially related to predicting the missing data. In addition, in order to include other auxiliary covariates in the imputations that are potentially related to missingness, logistic regression will be performed with the dependent variable missing/not missing. Only imputed values of independent variables will be used in the analyses. Multiple imputation will be performed with the R package mi.

The data being collected from the patient journals are to be used to monitor compliance with antibiotic use, kefir consumption, and any symptoms of C. diff infection. These data will be particularly useful in the event that there is no difference seen in C. diff infection rates among the study groups. From the self-reported patient data, compliance can be monitored and exclusion from the study may be warranted in the case of non-compliance.

ELIGIBILITY:
Inclusion Criteria:

Patients who have:

* Been admitted to the medical unit on 7 West at St. Luke's Hospital (Duluth, MN)
* Been prescribed a systemic antibiotic of any kind (administered by oral or parenteral route), but have not yet started the regimen
* Consented to be randomized and take part in the study and are adults greater than 19 years of age

Exclusion Criteria:

Patients who are/have:

* Tube feeding
* Undergoing dialysis and other renal treatment
* An existing C. difficile infection
* A recent history of C. difficile infection (within the last 3 months)
* A recent history of antibiotic use (within the last 3 months)
* Inflammatory bowel disease, Crohn's disease, or other chronic gastrointestinal syndrome
* A history of acquired of genetic immunodeficiencies; active, acute or chronic serious infections (i.e., viral hepatitis, HIV/AIDS), or autoimmune disorders
* Undergoing gastrointestinal surgery, radiation, or cytotoxic chemotherapy
* Allergy to milk protein

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-11; Primary Completion 2019-05-10 (Actual); Study Completion 2019-05-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johan S Bakken, M.D., Ph.D., Principal Investigator — St. Luke's Hospital of Duluth

REFERENCES:
- [Background] Zilberberg MD, Shorr AF, Kollef MH. Increase in adult Clostridium difficile-related hospitalizations and case-fatality rate, United States, 2000-2005. Emerg Infect Dis. 2008 Jun;14(6):929-31. doi: 10.3201/eid1406.071447. PMID 18507904
- [Background] Gerding DN, Muto CA, Owens RC Jr. Treatment of Clostridium difficile infection. Clin Infect Dis. 2008 Jan 15;46 Suppl 1:S32-42. doi: 10.1086/521860. PMID 18177219
- [Background] Lo Vecchio A, Cohen MB. Fecal microbiota transplantation for Clostridium difficile infection: benefits and barriers. Curr Opin Gastroenterol. 2014 Jan;30(1):47-53. doi: 10.1097/MOG.0000000000000023. PMID 24275671
- [Background] Bakken JS. Staggered and tapered antibiotic withdrawal with administration of kefir for recurrent Clostridium difficile infection. Clin Infect Dis. 2014 Sep 15;59(6):858-61. doi: 10.1093/cid/ciu429. Epub 2014 Jun 9. PMID 24917658
- [Background] Bakken JS. Resolution of recurrent Clostridium difficile-associated diarrhea using staggered antibiotic withdrawal and kefir. Minn Med. 2009 Jul;92(7):38-40. PMID 19708314
- [Background] Goldenberg JZ, Ma SS, Saxton JD, Martzen MR, Vandvik PO, Thorlund K, Guyatt GH, Johnston BC. Probiotics for the prevention of Clostridium difficile-associated diarrhea in adults and children. Cochrane Database Syst Rev. 2013 May 31;(5):CD006095. doi: 10.1002/14651858.CD006095.pub3. PMID 23728658
- [Background] Bolla PA, Carasi P, Bolla Mde L, De Antoni GL, Serradell Mde L. Protective effect of a mixture of kefir-isolated lactic acid bacteria and yeasts in a hamster model of Clostridium difficile infection. Anaerobe. 2013 Jun;21:28-33. doi: 10.1016/j.anaerobe.2013.03.010. Epub 2013 Mar 29. PMID 23542116
- [Background] Cohen SH, Gerding DN, Johnson S, Kelly CP, Loo VG, McDonald LC, Pepin J, Wilcox MH; Society for Healthcare Epidemiology of America; Infectious Diseases Society of America. Clinical practice guidelines for Clostridium difficile infection in adults: 2010 update by the society for healthcare epidemiology of America (SHEA) and the infectious diseases society of America (IDSA). Infect Control Hosp Epidemiol. 2010 May;31(5):431-55. doi: 10.1086/651706. PMID 20307191
- [Background] Su, Yu-Sung, et al.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The objective is to identify a population of at-risk patients that are undergoing treatment at St. Luke's Hospital (Duluth, MN) and CHI Creighton University Medical Center (Omaha, NE). The study will include patients who have been prescribed a systemic antibiotic of any kind (administered by oral or parenteral route), but have not yet begun the treatment regimen.
Pre-assignment Details: None, participants are randomized prior to any study activities
Period: Overall Study
Arm/Group | Group A | Group B | Group C
Started | 2 | 0 | 0
Completed | 2 | 0 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: There was not a sufficient patient population that qualified to participate in the study at our site
Groups:
- Total: Total of all reporting groups
Arm/Group | Group A | Group B | Group C | Total
Number analyzed (Participants) | 2 | 0 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants] — Population: There was not a sufficient patient population that qualified to participate in the study at our site.
  Participants
    <=18 years | 0 |  |  | 0
    Between 18 and 65 years | 2 |  |  | 2
    >=65 years | 0 |  |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 0 | 1
  Male | 1 | 0 | 0 | 1
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Diarrhea Among the Three Randomized Study Groups Over Time
Description: The overall incidence of diarrhea, represented as a percentage of patients, that develop diarrhea during the course of their enrollment in the study (an average of 35 days).
Time Frame: Assessed daily during hospitalization and daily for up to 30 days post-discharge; data will be represented as an overall incidence of diarrhea for all compliant patients upon study completion (average tracking time per patient is 35 days).
Population: Insufficient number of eligible participants enrolled and data were not collected
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Incidence of Clostridium Difficile Infection Among the Three Randomized Study Groups Over Time
Description: The overall incidence of C. difficile infections, represented as a percentage of patients, that develop diarrhea during the course of their enrollment in the study (an average of 35 days).
Time Frame: Assessed at any point during a patient's enrollment in the study (average of 35 days) when clinical symptoms require a C. difficile test per standard of care. Individual patients are tracked for an average of 35 days; data reported at study completion
Population: Insufficient number of eligible participants enrolled and data were not collected
Arm/Group | Group A | Group B | Group C
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 30 days
Description: Definitions do not differ from those provided by clinicaltrials.gov
Arm/Group | Group A | Group B | Group C
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-21): https://cdn.clinicaltrials.gov/large-docs/98/NCT02707198/Prot_SAP_000.pdf